CLINICAL TRIAL: NCT05734365
Title: Epidemiological, Clinical and Biological Characteristics and Therapeutic Management of ICU Patients With Severe Acute Exacerbation of COPD. Evaluation of the Prognosis and the Factors Associated With Survival Multicentre Prospective Observational Register
Brief Title: COPD-ICU Multicentre Prospective Observational Register
Acronym: COPD-ICU
Status: Recruiting | Type: Observational
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Alexis FERRE, Medical doctor, Principal investigator, Versailles Hospital
Other Study IDs: P 22/13
Record Dates: First submitted 2023-01-28; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: COPD Exacerbation Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COPD is one of the leading causes of morbidity, mortality and health care utilisation worldwide. Currently, COPD is the third leading cause of death worldwide and is therefore a major public health problem. Projections show an increase in the prevalence and burden of COPD in the coming decades due to ageing populations and continued exposure to risk factors.

In patients with COPD, mortality due to exacerbations is about 35%. Exacerbations represent the most important respiratory event in the history of this chronic disease and are of major socio-economic interest (about 50-75% of healthcare expenditure in this disease).

In the most severe cases, COPD exacerbations lead to respiratory distress with hypercapnic ventilatory acidosis requiring ventilatory support. These most severe episodes are common, accounting for 20% of exacerbations and are a signal of advanced disease, with a high risk of future hospitalisations and a limited long-term prognosis.

Despite progress in management, the mortality of these severe acute exacerbations is around 15% in the ICU and 20% in hospital. The long-term prognosis following hospitalisation for an acute exacerbation of COPD is poor with a 5-year mortality of around 50%. On the one hand, the means and treatments likely to improve the prognosis of these patients are of great medical and socio-economic interest, on the other hand, it seems important to identify the elements that may be associated with management failure and to treat them where appropriate.

Thus, improving scientific knowledge thanks to prospective data, evaluating the different characteristics and prognosis of patients hospitalised for a severe acute exacerbation of COPD seems, in the 21st century, a major axis in order to continue to optimise the individual management of these patients but also collectively, given the COPD public health burden.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years old
2. COPD documented or strongly suspected

   * Chronic respiratory symptoms (dyspnoea, cough and/or sputum)
   * Exposure to a known risk factor for COPD (such as tobacco smoke)
   * If available, respiratory function tests showing non- or partially reversible obstructive syndrome (post-bronchodilator ratio FEV1/CV < 0.7)
3. Severe acute exacerbation, defined as a worsening of the patient's usual respiratory symptoms with signs of acute respiratory distress (polypnoea ≥ 30 cycles.min-1 or use of accessory respiratory muscles) and/or hypercapnic acidosis (with PaCO2 ≥ 45 mmHg and pH ≤ 7.35)
4. Admission to an ICU, or a dedicated respiratory intensive care unit

Exclusion Criteria:

1. Known asthma (according to the criteria of the international "Global Initiative for Asthma" guidelines)
2. Patient refusal to participate (information note, application for non-opposition)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU, a step-unit or respiratory care unit for a severe acute exacerbation of COPD
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ICU survival | immediately after hospitalization in ICU
  vital status at ICU discharge
Day 90 survival | 90 days after ICU admission
  vital status at day 90

SECONDARY OUTCOMES:
One-year survival | one year after ICU admission
  Rate of survivors and non-survivors will be assessed at one year
  To better understand the one-year survival outcome, numerous factors will be assessed for an association with one-year survival: Demographic characteristics and chronic comorbidities; COPD severity; performans status; chronic use of long term oxygen therapy, systemic steroids or homecare non-invasive ventilation; previous intubation for COPD exacerbation; type of triggering factors of COPD exacerbation; type of treatment used during ICU stay (systemic steroids, intravenous bronchodilators, non-invasive ventilation and invasive ventilation); decision of withholding and withdrawal of care during ICU and hospital stay; further COPD exacerbation between hospital discharge and one year outcome; further COPD exacerbation requiring hospitalization between hospital discharge and one year outcome.
  We will perform descriptive analysis and multivariate analysis with odds ratio for each factor
Factors associated with ICU mortality | immediately after hospitalization in ICU
  Numerous factors will be assessed for an association with ICU mortality: Demographic characteristics and chronic comorbidities; COPD severity; performans status; chronic use of long term oxygen therapy, systemic steroids or homecare non-invasive ventilation; previous intubation for COPD exacerbation; type of triggering factors of COPD exacerbation; vital parameters at ICU admission (temperature, heart rate, mean arterial pressure, respiratory rate, coma glasgow scale); SAPS 2; arterial blood gaz results prameters at ICU admission; biological sample results at ICU admission; type of treatment used during ICU stay (systemic steroids, intravenous bronchodilators, non-invasive ventilation and invasive ventilation).
  We will perform descriptive analysis and multivariate analysis with odds ratio for each factor
Factors associated with hospital mortality | immediately after hospital discharge
  Numerous factors will be assessed for an association with hospital mortality: Demographic characteristics and chronic comorbidities; COPD severity; performans status; chronic use of long term oxygen therapy, systemic steroids or homecare non-invasive ventilation; previous intubation for COPD exacerbation; type of triggering factors of COPD exacerbation; vital parameters at ICU admission (temperature, heart rate, mean arterial pressure, respiratory rate, coma glasgow scale); SAPS 2; arterial blood gaz results prameters at ICU admission; biological sample results at ICU admission; type of treatment used during ICU stay (systemic steroids, intravenous bronchodilators, non-invasive ventilation and invasive ventilation).
  We will perform descriptive analysis and multivariate analysis with odds ratio for each factor
Factors associated with the need for invasive mechanical ventilation | immediately after the intervention named invasive mechanical ventilation
  Numerous factors will be assessed for an association with invasive mechanical ventlation: Demographic characteristics and chronic comorbidities; COPD severity; performans status; chronic use of long term oxygen therapy, systemic steroids or homecare non-invasive ventilation; previous intubation for COPD exacerbation; type of triggering factors of COPD exacerbation; vital parameters at ICU admission (temperature, heart rate, mean arterial pressure, respiratory rate, coma glasgow scale); SAPS 2; arterial blood gaz results prameters at ICU admission; biological sample results at ICU admission; type of treatment before ICU admission (systemic steroids, non-invasive ventilation) and type of treatment used during ICU stay (systemic steroids, intravenous bronchodilators, non-invasive ventilation).
  We will perform descriptive analysis and multivariate analysis with odds ratio for each factor

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ferré, MD, Principal Investigator — Centre hospitalier de Versailles, 78150, Le Chesnay
Locations (1):
- Centre hospitalier de Versailles, Le Chesnay, France